CLINICAL TRIAL: NCT03589716
Title: Evaluating the Accuracy of an Integrated Vital Sign Measurement Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Vital USA, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018P000152
Record Dates: First submitted 2018-06-04; First posted 2018-07-18 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Multimorbidity
Keywords: Vital Signs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Vital Signs Within Normal Range (Other): All participants will be asked to have an arm and finger measurement conducted and undergo vital sign measurements using the Vital Moto Mod and reference devices for blood pressure, heart rate, respiration rate, blood oxygen saturation, and temperature. Participants with vital signs within the normal physiological range will also be asked to perform an optional exercise testing and/or undergo arterial blood gas measurement.
  Interventions: Other: Vital Moto Mod; Other: Welch Allyn Connex Spot Vital Signs Monitor; Other: Capnostream 20 Portable Bedside Capnograph; Other: Welch Allyn 767 Mobile Aneroid Sphygmomanometerand 3M Littmann Master Classic II Teaching Stethoscope; Other: Scifit 1000R cycle ergometer
- Participants with Vital Signs Outside of Normal Range (Other): All participants will be asked to have an arm and finger measurement conducted and undergo vital sign measurements using the Vital Moto Mod and reference devices for blood pressure, heart rate, respiration rate, blood oxygen saturation, and temperature. Participants with vital signs outside of the normal physiological range would be documented.
  Interventions: Other: Vital Moto Mod; Other: Welch Allyn Connex Spot Vital Signs Monitor; Other: Capnostream 20 Portable Bedside Capnograph; Other: Welch Allyn 767 Mobile Aneroid Sphygmomanometerand 3M Littmann Master Classic II Teaching Stethoscope

INTERVENTIONS:
Other: Vital Moto Mod — All participants receive vital signs measurement using the Vital Moto Mod device and reference devices. The vital signs measured are blood pressure, heart rate, respiratory rate, oxygen saturation and temperature.
Other: Welch Allyn Connex Spot Vital Signs Monitor — This is the FDA approved reference device to measure heart rate, SpO2 and temperature.
Other: Capnostream 20 Portable Bedside Capnograph — This is the reference device to be used to obtain etCO2 waveforms for respiratory rate assessment.
Other: Welch Allyn 767 Mobile Aneroid Sphygmomanometerand 3M Littmann Master Classic II Teaching Stethoscope — These reference devices will be used together for blood pressure measurements.
Other: Scifit 1000R cycle ergometer — This is the device that will be used for exercise testing
  Arms: Participants with Vital Signs Within Normal Range

SUMMARY:
Partners Connected Health will conduct a clinical validation study to evaluate the accuracy of measurement for each vital sign with the Vital Moto Mod platform, compared to appropriate reference devices used in the hospital setting. The study will recruit volunteers from the Partners Healthcare network of clinics and hospitals and the general public.

DETAILED DESCRIPTION:
To assess the comparative clinical performance of the Vital Moto Mod device in the measurement of five vital signs (body temperature, respiratory rate, heart rate, oxygen saturation and blood pressure) in correlation with a reference device used in the hospital environment for vital sign measurement.

Vital sign measurement is a core process in delivering healthcare. Body temperature, respiratory rate, heart rate, oxygen saturation and blood pressure are some of the most frequently measured vital signs in inpatient as well as outpatient encounters. Currently, separate devices exist for measurement of each of these vital signs, each of which may have to be measured several times in a day. Consequently, measurement of vital signs is a time and human resource intensive process. Moreover, most of the devices currently used to measure vital signs cannot transmit data to the electronic medical record of patient, thereby creating opportunities for human error. VVVital USA has used proprietary sensor technology to develop Vital Moto Mod - a vital sign measurement platform that can non-invasively measure body temperature, respiratory rate, heart rate, oxygen saturation and blood pressure from a person's index finger, and allows this information to be pushed into their electronic medical/health record from the point of care

The primary market focus use of the Vital Moto Mod is to replace the vital sign cart in hospitals. Vital sign carts are expensive and cumbersome to move around the hospital. At a fraction of the cost, the Vital Moto Mod provides the same functionality including bar code scanning at a fraction of the cost. Additionally, the Vital Moto Mod can also be used at home without the need for a trained nurse. The Vital Moto Mod App will guide a user through the workflow of performing the measurements. The Vital Moto Mod is connected to a smartphone for storage, and has a USB interface for charging, thereby requiring no electrical connections during use. All measurements are taken by the device independent of the phone.

Partners Connected Health will conduct a clinical validation study to evaluate the accuracy of measurement for each vital sign with the Vital Moto Mod platform, compared to appropriate reference devices used in the hospital setting. The study will recruit volunteers from the Partners Healthcare network of clinics and hospitals and the general public.

ELIGIBILITY:
Inclusion Criteria:

For volunteers with one or more vital signs presumed to be within normal physiological range, at rest:

* Age ≥ 18 years
* Willing to allow arm and finger size to be measured
* Willing to allow measurement of skin color (optional)a
* Willing to undergo exercise testing (optional);
* Willing to allow an arterial blood gas draw (optional);

For volunteers with one or more vital signs expected to be outside of normal physiological range, at rest:

* Age≥18 years
* Willing to allow arm and finger size to be measured
* Willing to allow measurement of skin color (optional)

Exclusion Criteria:

For Volunteers Undergoing Heart Rate and Oxygen Saturation Measurement:

* Nail paint or artificial nail on the index finger of the left hand
* SpO2 less than 94%

For Volunteers Undergoing Exercise Testing with Vital Signs within Normal Physiological Range, at rest:

* Volunteers with vital signs outside of normal physiological range (ascertained during measurements conducted at study site before exercise testing)
* Age 65 years or older
* Consumption of food, alcohol or caffeine (coffee, tea or caffeinated soft-drinks) in a 3-hour period prior to testing
* Uncomfortable clothing, or inappropriate footwear for exercise testing
* Self-report of any of the following:
* History of fall or fracture in the past year
* History of arthritis
* History of dizziness
* History of neurological illness
* History of chest pain or myocardial infarction
* History of hypertension or diabetes mellitus
* History of heart disease
* History of stroke or transient ischemic attack
* Active treatment for anemia, electrolyte imbalance, or hyperthyroidism
* Physical disability that precludes safe and adequate testing
* Mental impairment with limited ability to cooperate4
* Pregnancy (Volunteer will be excluded if either of the following is true: a) self-report of being pregnant; b) positive urine pregnancy test)

For Volunteers undergoing an Arterial Blood Gas Draw with Vital Signs within Normal Physiological Range, at rest:

* Self-reported history of a clotting disorder of the blood, or active treatment with medicines affecting blood clotting (e.g. Warfarin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of Vital Moto Mod vital signs measurements in agreement with reference device vital signs measurements | 1 day
  Vital signs measurements for each participant would be compared using the Vital Moto Mod and reference devices for blood pressure, heart rate, respiratory rate, oxygen saturation and temperature

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Partners Connected Health, Boston, Massachusetts, United States